CLINICAL TRIAL: NCT01641354
Title: Reversible Hemiepiphysiodesis in Children - Stapling Versus Eight Plate
Brief Title: Comparison of Two Surgical Techniques to Treat Knock Knees in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Martin Gottliebsen, PhD-student, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-20080179; J.nr. 2009-41-3248 (Other: Datatilsynet)
Record Dates: First submitted 2010-06-07; First posted 2012-07-16 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Genu Valgus
Keywords: Hemiepiphysiodesis
MeSH Terms: conditions — Genu Valgum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Hemiepiphysiodesis — Partial closure of growth plate to correct deformity

SUMMARY:
Knock knees or genu valgus necessitates in some children corrective surgery with partial closure of the growth plate at level of the knee.

DETAILED DESCRIPTION:
Background: Genu valgus is a condition with malalignment of the lower extremity. Surgery may be indicated in severe cases and reversible hemiepiphysiodesis is often the treatment of choice in growing children. Partial closure can be obtained by stapling technique or with a new treatment called tension band plating.

ELIGIBILITY:
Inclusion Criteria:

* genu valgus
* remaining growth

Exclusion Criteria:

* systemic disease
* unilateral disease

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-07 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Treatment time | up to 3 years

SECONDARY OUTCOMES:
Pain score post operatively | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Gottliebsen M, Rahbek O, Hvid I, Davidsen M, Hellfritzsch MB, Moller-Madsen B. Hemiepiphysiodesis: similar treatment time for tension-band plating and for stapling: a randomized clinical trial on guided growth for idiopathic genu valgum. Acta Orthop. 2013 Apr;84(2):202-6. doi: 10.3109/17453674.2013.782526. Epub 2013 Mar 14. PMID 23485073